CLINICAL TRIAL: NCT00584597
Title: The Safety and Efficacy of the Homeopathic Medication TRAUMEEL S for the Treatment of Radiation-Induced Mucositis
Brief Title: A Trial of Homeopathic Medication TRAUMEEL S for the Treatment of Radiation-Induced Mucositis
Acronym: TRAUMEEL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Greg Krempl, MD, University of Oklahoma Health Sciences Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TRAUMEEL_S_Krempl
Record Dates: First submitted 2007-12-20; First posted 2008-01-02 (Estimated); Last update posted 2010-12-13 (Estimated); Status verified 2010-12

CONDITIONS: Mucositis; Head and Neck Cancer
Keywords: Radiation-Induced Mucositis; Head and neck cancer; TRAUMEEL; Mucositis; Radiation; Oral cancer; Inflammation of the mouth; Homeopathic Medication
MeSH Terms: conditions — Mucositis; Head and Neck Neoplasms; Mouth Neoplasms; Stomatitis | interventions — Sodium Chloride; Traumeel S

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Placebo Comparator): Saline
  Interventions: Drug: Saline
- 2 (Experimental): Traumeel S 1 mL
  Interventions: Drug: Traumeel S
- 3 (Experimental): Traumeel S 2 mL
  Interventions: Drug: Traumeel S
- 4 (Experimental): Traumeel S 3 mL
  Interventions: Drug: Traumeel S

INTERVENTIONS:
Drug: Saline — Saline Control
  Arms: 1
Drug: Traumeel S — Traumeel S 1 mL
  Arms: 2
Drug: Traumeel S — Traumeel S 2mL
  Arms: 3
Drug: Traumeel S — Traumeel S 3mL
  Arms: 4

SUMMARY:
The specific aim of this study will be to determine the safety of TRAUMEEL S for mucositis in head and neck cancer patients undergoing radiation therapy.

DETAILED DESCRIPTION:
Oral mucositis is a debilitating side effect of radiation therapy for head and neck cancer patients. The severe inflammation of the oral cavity can be detrimental to quality of life and cause interruption in vital cancer treatment. Despite numerous proposed therapies, an effective agent for oral mucositis has yet to be found. TRAUMEEL S, a homeopathic remedy made up of highly diluted botanical extracts and minerals, has shown benefit for mucositis in children undergoing chemotherapy. The objective of this study is to evaluate the safety of TRAUMMEL S in the prevention and treatment of radiation-induced oral mucositis. The patients will use the medication as a mouthwash during radiation therapy and will be evaluated weekly with physical examination criteria and questionnaires for symptoms and side effects.

ELIGIBILITY:
Inclusion Criteria:

* Head and neck cancer patients post resection of primary tumor with negative or microscopically positive surgical margins
* Patients undergoing planned radiation therapy
* Age 18 to 99
* Nonsmokers

Exclusion Criteria:

* Head and neck cancer patients post resection of primary tumor with grossly positive surgical margins
* Patients receiving adjuvant chemotherapy
* Pediatric patients (age < 18)
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2005-10; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
The specific aim will be to determine the safety of TRAUMEEL S for mucositis in head and neck cancer patients undergoing radiation therapy | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Greg Krempl, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States